CLINICAL TRIAL: NCT05609305
Title: FAcilitating Safe Transition to Home for Preterm Infants: an Observational Study
Acronym: FAST-Home
Status: Active, not recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 314885
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-11

CONDITIONS: Infant, Premature, Discharge
MeSH Terms: conditions — Premature Birth | interventions — Drainage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Discharge — observational study, not intervention

SUMMARY:
Finding out what the common discharge barriers are in neonatal units will help design and develop services to facilitate safe, early discharge in preterm babies. This study will have 2 components. Retrospectively the study team will study the electronic medical records of preterm infants admitted to 20 neonatal units throughout the UK to identify the PMA at which each of the barriers to discharge are reached and identify the final discharge barrier. In a smaller-scale prospective study, the study team will investigate what is the final discharge barrier for infants admitted for neonatal care in the Royal Derby Hospital. The study team will follow up with the family, 2 weeks after discharge home, to find out if the infant has remained well and not required readmission to the hospital (information which will not be available in the electronic patient records analysed retrospectively). This will help determine whether the discharge was appropriate and safe.

DETAILED DESCRIPTION:
Infants born before 37 completed weeks of gestation are expected to need additional care and are routinely admitted to neonatal units in the UK. Neonatal care in the National Health Service (NHS) is designated as intensive or high dependency care when infants need intensive support such as with breathing (e.g., mechanical ventilation), nutrition (e.g., parenteral nutrition) and/or other medical needs (e.g., cardiovascular support with inotropes). With increasing maturity, preterm infants stop needing these and spend some time with less additional support such as for feeding and keeping warm while they grow and mature sufficiently to go home safely. This period is designated as "special care."

Depending on how premature babies are and other medical needs, preterm infants spend a varying length of time in the hospital with most going home between 37 and 40 weeks post-menstrual age (PMA)1. PMA is the time elapsed between the first day of the mother's last menstrual period (as a marker of the day when the pregnancy started) and the current age. Length of hospital stay (number of days from birth to discharge home) and PMA at discharge are inversely correlated with gestational age at birth i.e., the more premature the infant, the longer they stay in hospital and the more likely they are to be at a higher PMA when going home. Data from the National Neonatal Research Database (NNRD), which collects information from all NHS neonatal units in the UK, showed that, between 2011 and 2014, infants born at 24 weeks' GA spent an average of 123 days in the hospital (going home at the average PMA of 41.6 weeks) which reduced to an average of 34 days (and PMA 35.9 weeks) for those born at 31 weeks' GA. With more recent data (2010-2020), we found that infants born at 22-26 weeks' GA have a length of the hospital (median (IQR)) of 88 (69-110) days while those born at 27-31 weeks' stay for 44 (33-57) days. The more immature group (22-26 weeks' GA) were 38 (36-41) weeks' PMA at discharge while 27-31 weeks' infants were 36 (35-37) PMA at discharge (Szatkowski et al., unpublished). These data show that preterm infants need a considerable period to get ready to be discharged home.

Although neonatal care is lifesaving and its availability has, undoubtedly, improved the survival and well-being of premature infants; staying in the neonatal unit longer than necessary can be detrimental to the preterm infant and family. The environment of neonatal units with bright lights, noise, and lack of one-to-one developmental care can have adverse effects on the infant's development. Prolonged hospitalisation also means prolonged separation from the family and continued stress for parents. In parent and public consultation during the set-up of the FEED1 trial, a large, ongoing randomised controlled trial in the UK, it was found that parents overwhelmingly supported the need to find ways to reduce the length of hospital stay. The parents said that reducing the time spent in the hospital "by even a few days" would improve their well-being significantly.

Prolonged hospitalisation also means an increased cost of care. A reduction in length of stay can save money for the NHS. The 2020/21 tariff for NHS care specifies the cost of care for infants in neonatal units. The cost of one day of "special care" is £709.16 (https://www.england.nhs.uk/costing-in-the-nhs/national-cost-collection/). From 2012-2020, there were, on average, approximately 39,000 infants born each year before 37 weeks' GA cared for in neonatal units in the UK6. If, with a better understanding of discharge barriers and optimal discharge planning, length of stay could be reduced by 2 days per infant, the NHS would save approximately £56 million per year.

Earlier discharge is safe and improves parental well-being and quality of life at home and can save millions of pounds in cost of care. However, before a preterm infant can go home, it must be ensured that infants are ready to be discharged safely.

A comprehensive, well-planned discharge of a medically stable infant helps ensure a positive transition to home and safe, and effective care after discharge. "Discharge readiness" of a preterm infant typically requires a level of physiological maturity such that the infant can:

Maintain body temperature: in the initial days after birth, most preterm infants are nursed in incubators. As their ability to generate heat and maintain body temperature matures, they spend some time in heated cots and are finally moved into regular baby cots with normal clothing and blankets as they would have at home.

Breathe on their own: preterm babies have immature lungs and often also have long pauses in their breathing (apnoea of prematurity). Many require breathing support and caffeine to help them breathe effectively and regularly. As breathing ability and control mature, infants can breathe on their own without significant pauses. Some may continue to need additional oxygen and may go home on home oxygen therapy.

Feed adequately: Preterm infants take time to establish feeding. Initially, they may need parenteral nutrition. Milk feeds are slowly introduced via a gastric tube. As their ability to suck and swallow matures, infants learn to feed orally. This can be on the mother's breast or taking the mother's milk or infant formula milk by a bottle. Infants with significant respiratory issues or other co-morbidities may take longer to establish oral feeding. To be safely discharged home, infants should be able to take their milk requirements orally. Occasionally, where the service is available, infants who can take most of their milk orally can be safely discharged home with partial gastric feeding.

Gain weight: Milk intake in preterm infants should be sufficient to support adequate weight gain. Most infants are considered ready to be discharged home if they are at least 1700-1800g in weight and gaining weight on their regular feeding regimen.

In addition to these, neonatal teams must ensure that the family and home are prepared to assume care of the preterm infant. This includes basic care such as keeping warm, feeding, bathing, safe travel, and other needs such as giving medicines. The family's emotional readiness and confidence are equally important. Neonatal units provide a package of support for getting parents ready to take their baby home.

Most infants reach the level of maturity required for safe discharge at a variable pace and may become mature in one aspect but not the others e.g., an infant may be able to breathe well, maintain temperature, and be gaining weight, but is unable to take sufficient oral feeds. In this case, the reason the infant needs to stay in the hospital longer becomes their inability to feed orally. This is referred to as the infant's "terminal or final discharge barrier" i.e., the aspect of physiological maturity that is the reason to stay in the hospital for longer. There is very little research to investigate the barriers to safe discharge home and information on what the most common "final discharge barrier" is in the UK population of preterm infants. This information will help us identify and target areas where we can design and evaluate future quality improvement and other approaches to enable sooner and safer discharge. In a study in the USA, the team at the neonatal unit in Birmingham, Alabama found that independent oral feeding was the main final discharge barrier in their unit. They planned and implemented a quality improvement project to support independent oral feeding and reduced the length of hospital stay by 1 week.

Finding out what the common discharge barriers are in neonatal units will help us design and develop services to facilitate safe, early discharge in preterm babies. This study will have 2 components. Retrospectively the study team will study the electronic medical records of preterm infants admitted to 20 neonatal units throughout the UK to identify the PMA at which each of the barriers to discharge are reached and identify the final discharge barrier. In a smaller-scale prospective study, the study team will investigate what is the final discharge barrier for infants admitted for neonatal care in the Royal Derby Hospital. The study team will follow up with the family, 2 weeks after discharge home, to find out if the infant has remained well and has not required readmission to the hospital (information which will not be available in the electronic patient records analysed retrospectively). This will help the study team determine whether the discharge was appropriate and safe.

ELIGIBILITY:
Inclusion Criteria:

* Born at <37 weeks' gestational age (GA)
* Admitted to neonatal care for >48 hours
* Discharged home alive

For prospective component:

*Parent or legal guardian available who can give informed consent

Exclusion Criteria:

* Infants with major congenital anomalies or genetic syndromes
* Infants who die before discharge home
* Infants who are transferred for continuing care outside of neonatal service before discharge home

Ages: 26 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All admissions from 01/01/2012 to 31/12/22 to NICU <37 weeks
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Final barrier to discharge home | 01/01/2012 to 31/12/22
  defined as the last to be achieved
  Able to maintain thermoregulation without additional support
  Breathing spontaneously without any caffeine (without supplemental oxygen or in supplemental oxygen (<1L/min) with plan for home oxygen therapy) without any episodes of apnoea for at least 5 days
  Achieved safe oral feeding (adequate oral feeds or are ready for discharge on home NG-feeding regimen)
  defined as the last of the following four to be achieved, Able to maintain thermoregulation without additional support
  Breathing spontaneously without any caffeine (without supplemental oxygen or in supplemental oxygen (<1L/min) with plan for home oxygen therapy) without any episodes of apnoea for at least 5 days
  Achieved safe oral feeding (adequate oral feeds or are ready for discharge on home NG-feeding regimen)
  Achieved a weight of at least 1700 grams

SECONDARY OUTCOMES:
age | 01/01/2012 to 31/12/22
  age on discharge

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Derby and Burton, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan